CLINICAL TRIAL: NCT00914264
Title: The Continuous Positive Airway Pressure Effects on Chronic Obstructive Pulmonary Disease Patients With Obstructive Sleep Apnea
Brief Title: The Effects of Continuous Positive Airway Pressure on Overlap Syndrome
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 972246B
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2010-08

CONDITIONS: COPD & OSA
Keywords: chronic obstructive airway disease; obstructive sleep apnea; continuous positive airway pressure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- COPD with OSA with CPAP treatment: COPD with OSA: CPAP treatment
  Interventions: Device: continuous positive airway pressure
- COPD without OSA: COPD without OSA, not treat with CPAP
- COPD with OSA but without CPAP treatment: COPD with OSA but patient refused CPAP treatment

INTERVENTIONS:
Device: continuous positive airway pressure — CPAP with adequate pressure for 1 day, 3 & 12 months
  Groups: COPD with OSA with CPAP treatment

SUMMARY:
1. The first objective of this study is to determine the differences between, while the airway obstruction severity is the same, and the acute continuous positive airway pressure (CPAP) effect on chronic obstructive pulmonary disease (COPD) patients with overlap syndrome compared with COPD patients without in terms of sleep quality, autonomic nerve activity, biologic markers of systemic inflammatory, and exercise performance.
2. The second objective of this study is to evaluate the subacute (3 months treatment) CPAP effect on COPD patients with overlap syndrome in terms of pulmonary hemodynamic and right heart function, We will also determine the subacute effect of CPAP on sleep and life quality, autonomic nerve activity, biologic markers of systemic inflammatory, as well as exercise performance.
3. The last objective of this study is to evaluate the long term (12 months treatment) CPAP effect on COPD patients with overlap syndrome. The un-scheduled clinic or emergency department visiting, hospitalization, or mortality will be recorded to see if there is significant treatment effect in terms of reducing morbidity and mortality. The long term CPAP effect on sleep and life quality, autonomic nerve activity, biologic markers of systemic inflammatory, exercise performance, as well as pulmonary hemodynamic and right heart function will be re-evaluation.

DETAILED DESCRIPTION:
COPD patients will be disturbed by season 12 months follow up is better than 18 months

ELIGIBILITY:
Inclusion Criteria:

* chronic stable COPD
* FEV1/FVC < 70%
* No response to beta-agonist
* without acute exacerbation within2 months

Exclusion Criteria:

* Chronic respiratory failure (PaO2<60 mmHg, PaCO2>50 mmHg)
* Clinical evidence of congestive heart failure
* Facial defect and all the other condition that can't tolerate nasal mask
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from outpatient clinic of CGMH and those in COPD cohort
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
exercise performance | 3 days, 3 & 12 months
  the condition of COPD patient will be disturbed by season factor 12 months follow up will be better than 18 months

SECONDARY OUTCOMES:
autonomic nerve activity | 3 days, 3 & 12 months
  the same reason as above
mortality and acute exacerbation | 1, 5, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Lun Lo, MD, Study Director — Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan; Tsai-Yu Wang, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan; Han-Pin Kuo, MD,PHD, Study Chair — Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan
Locations (1):
- Division of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang TY, Lo YL, Lee KY, Liu WT, Lin SM, Lin TY, Ni YL, Wang CY, Ho SC, Kuo HP. Nocturnal CPAP improves walking capacity in COPD patients with obstructive sleep apnoea. Respir Res. 2013 Jun 19;14(1):66. doi: 10.1186/1465-9921-14-66. PMID 23782492